CLINICAL TRIAL: NCT04631250
Title: A Split-Face Clinical Trial of Conventional Photodynamic Therapy Versus Daylight Photodynamic Therapy for The Treatment of Acne Vulgaris
Brief Title: Conventional Photodynamic Therapy Versus Daylight Photodynamic Therapy for The Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0043-18
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; photodynamic therapy; PDT; Daylight PDT
MeSH Terms: conditions — Acne Vulgaris | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: "Split Face design" is a common model used in dermatology to study the difference between two treatments on a facial condition. The face was divided into two symmetrical contralateral treatment areas: the left was covered with a light-impermeable dressing, while the right face was exposed to sunlight. After 2 hours outdoors, the right side of the face was covered, and the left half was illuminated with red light.
Who Masked: Outcomes Assessor
Masking Description: The photographs of the patients were evaluated by two dermatologists blinded to the study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Right: daylight illumination (Experimental): The right side of the face was treated using daylight PDT
  Interventions: Drug: 5-Aminolevulinic Acid-Containing Product in Cutaneous Dose Form
- Left face: conventional illumination with red light (Experimental): The left side was treated with conventional PDT.
  Interventions: Drug: 5-Aminolevulinic Acid-Containing Product in Cutaneous Dose Form

INTERVENTIONS:
Drug: 5-Aminolevulinic Acid-Containing Product in Cutaneous Dose Form — 5-Aminolevulinic Acid was applied to both sides of the face.

SUMMARY:
Photodynamic therapy (PDT) is considered an effective treatment for acne vulgaris. The study aims to determine whether treatment with daylight as an illumination source is as effective as conventional, red light illumination.

15 patients with acne vulgaris received 4 treatment sessions at three-week intervals. First, 5-aminolevulinic acid (ALA) was applied to the entire face. Then the face was divided into two symmetrical contralateral treatment areas: the left was covered with a light-impermeable dressing, while the right face was exposed to sunlight. After 2 hours outdoors, the right side of the face was covered, and the left half was illuminated with red light.

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is considered an effective treatment for acne vulgaris .One of the most important drawbacks of PDT is the pain during illumination.

It has been shown that daylight PDT is an effective treatment for actinic keratosis. In order to examine the efficacy of daylight PDT for acne vulgaris, we used a split-face design: the face was divided into two symmetrical contralateral treatment areas: the left was covered with a light-impermeable dressing, while the right face was exposed to daylight. After 2 hours outdoors, the right side of the face was covered, and the left half was illuminated with red light.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of acne vulgaris on the face
* Acne lesions include inflammatory papules/ pustules/ nodules and cysts , and non-inflammatory open and closed comedones.
* Acne refractory to conventional therapies
* Patients who are unable or do not want to take oral isotretinoin
* Patients who cannot tolerate isotretinoin

Exclusion Criteria:

* History of oral retinoid use within 12 months of study entry
* Systemic antibiotics within 6 month of study entry
* Topical acne treatment within 1 month of study entry
* Presence of any other skin disease that could interfere with the assessment of the acne, such as folliculitis or rosacea
* Presence of any other systemic disease that could affect the acne severity by its presence, such as polycystic ovarian syndrome, or by any medication prescribed for the treatment of the systemic diseases (retinoids, antibiotics).
* Pregnancy or intention to get pregnant
* lactating woman
* Porphyria
* Photosensitive dermatoses
* Allergy to any component of the photosensitizer compound
* Personal history of melanoma or dysplastic nevi
* A beard or other facial hair that might interfere with study assessments;

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Reduction in acne lesion counts and total acne severity score on both sides of the face | We measured the difference between the number of lesions in the first visit and the number of lesions in the follow up visit, 12 weeks after the last teatment
  Change in the number of inflammatory and non-inflammatory acne lesions
Difference in adverse effects between the two sides | After each of the 4 treatment sessions
  Difference in pain scores, erythema after each treatment, erosions and pustulosis

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel